CLINICAL TRIAL: NCT02275884
Title: Evaluation of Plasma Concentrations of Pharmacologically Active Constituents of Chocolate and Their Symptomatic Effects in Patients With Idiopathic Parkinson's Disease
Brief Title: Pharmacologically Active Constituents of Chocolate and Their Symptomatic Effects in Patients With Idiopathic Parkinson's Disease
Acronym: Choc-PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: University of Wuerzburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EK366112012
Record Dates: First submitted 2014-10-17; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Cacao; Biogenic amines; Xanthines; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases | interventions — Chocolate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dark chocolate (85% cocoa) (Active Comparator): Patients will initially receive 50 grams of dark chocolate (85% cocoa) b.i.d. for one week. Patients will then cross over to intake of 50 grams of white chocolate (0% cocoa) b.i.d. for another week.
  Interventions: Dietary Supplement: Dark chocolate (85% cocoa); Dietary Supplement: White chocolate (0% cocoa)
- White chocolate (0% cocoa) (Sham Comparator): Patients will initially receive 50 grams of white chocolate (0% cocoa) b.i.d. for one week. Patients will then cross over to intake of 50 grams of dark chocolate (85% cocoa) b.i.d. for another week.
  Interventions: Dietary Supplement: Dark chocolate (85% cocoa); Dietary Supplement: White chocolate (0% cocoa)

INTERVENTIONS:
Dietary Supplement: Dark chocolate (85% cocoa)
Dietary Supplement: White chocolate (0% cocoa)

SUMMARY:
This study evaluates plasma concentrations of pharmacologically active constituents of chocolate and their effects on motor and non-motor symptoms of Parkinson's disease. Following one week of abstinence from cocoa-containing products, patients with Parkinson's disease will be randomized to receive either dark or white chocolate. After one week of chocolate consumption, patients will then cross over to white or dark chocolate, respectively, and take the corresponding chocolate product for another week. Blood samples will be taken at baseline, week 1 and week 2 to examine plasma concentrations of pharmacologically active constituents of chocolate at all three timepoints. Moreover, patients will be clinically examined for motor and non-motor symptoms at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Female or male individuals aged 40 years and above
* Parkinson's Disease according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria
* Hoehn and Yahr stage I-III
* Minimum score of 16 points in the motor part of the Unified Parkinson Disease Rating Scale (UPDRS part III)
* Stable antiparkinsonian medication for at least 4 weeks prior to study inclusion
* Ability to provide informed consent

Exclusion Criteria:

* Clinical signs for a secondary or atypical Parkinsonian syndrome
* Treatment with any investigational medical product within 30 days prior to study inclusion
* Intake of chocolate or other cocoa-containing products within the last 7 days prior to study inclusion (patients can be re-screened after 7 days of abstinence from chocolate and other cocoa-containing products)
* Known intolerance or allergies against chocolate or other cocoa-containing products
* Diabetes mellitus and/or impaired glucose tolerance in the medical history
* Alcohol or drug abuse in the medical history
* Presence of levodopa-induced motor complications
* Other neurological, psychiatric or miscellaneous conditions that would significantly impair study participation, medical assessments or the consenting process

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change in plasma concentrations of pharmacologically active constituents of chocolate after one week consumption of dark chocolate in comparison to baseline and to one week consumption of white chocolate | 7 days
Change in the severity of motor and non-motor symptoms of PD after one week consumption of dark chocolate in comparison to baseline and to one week consumption of white chocolate | 7 days
  Changes in motor symptoms will be assessed with the UPDRS, changes in non-motor symptoms will be assessed with NMSS and NMSQuest.

SECONDARY OUTCOMES:
Change in cognitive measures (MoCA, SCOPA-COG) after one week consumption of dark chocolate in comparison to baseline and to one week consumption of white chocolate | 7 days
Change in depressive symptoms (BDI-II) after one week consumption of dark chocolate in comparison to baseline and to one week consumption of white chocolate | 7 days
Change in the quality of life (PDQ-39) after one week consumption of dark chocolate in comparison to baseline and to one week consumption of white chocolate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Löhle, MD, Principal Investigator — Department of Neurology, Dresden University of Technology
Locations (1):
- Department of Neurology, Dresden University of Technology, Dresden, Saxony, Germany